CLINICAL TRIAL: NCT01678586
Title: Effect of Acupuncture and Pain Medication on Radicular Pain Using QST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, M.D., Ph.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2012P-001795; 5R01AT005819-04 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: Pain; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Acupuncture Therapy; Gabapentin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- True Acupuncture (Active Comparator): Pain subjects with radicular pain receiving 6, 30 minute acupuncture treatments.
  Interventions: Other: Acupuncture
- Sham Acupuncture (Sham Comparator): Pain subjects with radicular pain receiving 6, 30 minute sham acupuncture treatments.
  Interventions: Other: Sham Acupuncture
- Gabapentin (Active Comparator): Pain subjects with radicular pain receiving gabapentin. Medication treatment groups will titrate up to the standard clinical treatment dosage for one week and maintain that dosage for 1.5 weeks.
  Interventions: Drug: Gabapentin
- Sham Gabapentin (Sham Comparator): Pain subjects with radicular pain receiving sham gabapentin. Medication treatment groups will titrate up to the standard clinical treatment dosage for one week and maintain that dosage for 1.5 weeks.
  Interventions: Drug: Sham Gabapentin

INTERVENTIONS:
Other: Acupuncture — In true acupuncture the needles penetrate the skin.
  Arms: True Acupuncture
Other: Sham Acupuncture — In sham acupuncture the needles do not penetrate the skin.
  Arms: Sham Acupuncture
Drug: Gabapentin — Gabapentin is a commonly prescribed drug used to treat neuropathic pain.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Sham Gabapentin — Benadryl or diphenhydramine is used as a placebo as it could mimic some common side effects of gabapentin (i.e. sedation, drowsiness, lightheadedness)
  Other Names: Benadryl, diphenhydramine
  Arms: Sham Gabapentin

SUMMARY:
In this aim, we propose to conduct a double blinded, placebo-controlled, and randomized clinical trial to compare the clinical effectiveness of radicular pain relief by either acupuncture therapy or a course of pain medication (e.g., Gabapentin) using Quantitative Sensory Testing (QST).

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between ages 18 to 75 years. Both male and female subjects will be recruited.
2. Subject should have had cervical or lumbar radicular pain for at least two months. This requirement is to avoid the uncertainty of an unstable pain condition and to minimize the study variation.
3. Subject has a pain score of 4 or above (visual analog scale, VAS: 0 - 10 from no pain to worst pain).
4. Cervical or lumbar radicular pain will include, but is not limited to, such clinical conditions as disk herniation, spinal stenosis, and post-laminectomy syndrome.

Exclusion Criteria:

1. Subject has detectable sensory deficits at the site of QST. Sensory deficits refer to such conditions resulting from neurological diseases or medical conditions causing peripheral polyneuropathy and sensory changes, which include but are not limited to diabetic neuropathy, alcoholic neuropathy, AIDS neuropathy, severe thyroid disease, and severe liver or kidney disorders.
2. Subject has scar tissue, infection, or acute injury at the site of QST.
3. Subject is pregnant.
4. Subject tests positive for illicit drugs.
5. Subject has a pacemaker.
6. Subject is currently taking gabapentin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chen L, Deng H, Houle T, Zhang Y, Ahmed S, Zhang W, Sullivan S, Opalacz A, Roth S, Filatava EJ, Stabach K, Vo T, Malarick C, Kim H, You Z, Shen S, Mao J. Comparison between acupuncture therapy and gabapentin for chronic pain: a pilot study. Acupunct Med. 2021 Dec;39(6):619-628. doi: 10.1177/09645284211026683. Epub 2021 Jul 29. PMID 34325532
- See also: Center for Translational Pain Research — https://www.massgeneral.org/anesthesia/translational-pain-research

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | True Acupuncture | Sham Acupuncture | Gabapentin | Sham Gabapentin
Started | 15 | 16 | 11 | 14
Completed | 14 | 15 | 9 | 12
Not Completed | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | True Acupuncture | Sham Acupuncture | Gabapentin | Sham Gabapentin | Total
Number analyzed (Participants) | 15 | 16 | 11 | 14 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 7 | 13 | 45
  >=65 years | 4 | 2 | 4 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (12.33) | 53.07 (9.28) | 54.89 (13.78) | 55.25 (6.08) | 54.66 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 6 | 7 | 29
  Male | 4 | 11 | 5 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 16 | 11 | 14 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 0 | 5 | 11
  White | 9 | 12 | 9 | 8 | 38
  More than one race | 0 | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 11 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Changes in QST Measures in Response to Acupuncture or Gabapentin at Visit 1, Visit 4 and Visit 7 for CS, WS, HP, CP (CS: Cold Sensation; WS: Warm Sensation; HP: Heat Pain; CP: Cold Pain)
Description: Changes in response to heat stimulation stated as pain, sensitivity and tolerance. Responses are measured with a quantitative sensory testing (QST) device. Measurements are taken before, during, and after acupuncture treatment and throughout the gabapentin medication regimen. Measurements are taken at Visit 1 (before any intervention), Visit 4 (after session 3 for acupuncture groups or within treatment week 2 for medication groups), and Visit 7 (after session 6 for acupuncture groups or within treatment week 3 for medication groups), up to a maximum of 3 weeks for each participant.
Time Frame: 3 weeks apart. Taken at Visit 1 (before any intervention), Visit 4 (after session 3 for acupuncture groups or within treatment week 2 for medication groups), and Visit 7 (after session 6 for acupuncture groups.
Population: Enrolled participants who didn't withdraw, were not withdrawn by the investigator.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | True Acupuncture | Sham Acupuncture | Gabapentin | Sham Gabapentin
Number analyzed (Participants) | 14 | 15 | 9 | 12
degree celsius
  Visit 1 Cold Sensation | 26.41 (5.01) | 26.54 (2.44) | 27.92 (2.22) | 24.25 (4.27)
  Visit 1 Warm Sensation | 38.43 (4.03) | 39.57 (4.63) | 38.49 (4.89) | 39.90 (4.61)
  Visit 1 Heat Pain | 45.77 (5.08) | 47.05 (3.55) | 46.31 (4.04) | 46.34 (4.33)
  Visit 1 Cold pain | 11.11 (11.77) | 8.20 (8.76) | 9.65 (10.87) | 9.87 (10.53)
  Visit 4 Cold Sensation | 26.04 (3.99) | 25.11 (6.73) | 28.38 (5.78) | 26.35 (3.90)
  Visit 4 Warm Sensation | 37.56 (3.91) | 39.15 (3.65) | 37.11 (3.45) | 37.50 (3.40)
  Visit 4 Heat Pain | 46.15 (3.46) | 47.51 (2.41) | 45.92 (4.07) | 45.34 (4.70)
  Visit 4 Cold Pain | 11.01 (10.22) | 9.55 (9.66) | 9.09 (9.89) | 14.13 (10.79)
  Visit 7 Cold | 26.17 (3.23) | 25.12 (2.10) | 27.04 (2.28) | 26.25 (3.96)
  Visit 7 Warm | 38.38 (4.34) | 39.09 (2.94) | 37.59 (3.64) | 38.33 (3.94)
  Visit 7 Heat Pain | 46.85 (2.96) | 47.69 (2.56) | 46.73 (1.91) | 44.64 (4.71)
  Visit 7 Cold Pain | 10.47 (8.87) | 8.42 (9.98) | 12.63 (10.05) | 13.82 (8.80)

2. Primary Outcome: Changes in QST Measures in Response to Acupuncture or Gabapentin at Visit 1, Visit 4 and Visit 7 HPT, CPT and Tol (HPT: Heat Pain Threshold; CPT: Cold Pain Threshold; Tol: Tolerance to 47°C Heat Stimulation)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Enrolled participants who didn't withdraw, were not withdrawn by the investigator.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | True Acupuncture | Sham Acupuncture | Gabapentin | Sham Gabapentin
Number analyzed (Participants) | 14 | 15 | 9 | 12
Seconds
  visit 1 heat pain threshold | 48.95 (2.86) | 49.93 (2.39) | 49.59 (2.49) | 48.95 (4.02)
  visit 1 cold pain threshold | 5.16 (6.78) | 4.7 (6.82) | 3.89 (8.58) | 6.8 (9.68)
  Visit 1 tolerance to 47 celsius heat simulation | 27.86 (25.39) | 27.56 (24.15) | 29.59 (28.43) | 23.63 (24.40)
  visit 4 heat pain threshold | 49.53 (1.96) | 50.39 (1.46) | 48.71 (2.91) | 48.55 (3.79)
  visit 4 cold pain threshold | 3.72 (6.95) | 2.1 (4.43) | 7.09 (8.53) | 7.05 (9.45)
  Visit 4 tolerance to 47 celsius heat simulation | 28.36 (26.67) | 29.1 (24.85) | 23.69 (26.44) | 25.23 (26.49)
  visit 7 heat pain threshold | 49.57 (2.39) | 50.34 (1.56) | 49.8 (2.01) | 48.40 (3.74)
  visit 7 cold pain threshold | 2.7 (4.36) | 2.38 (6.42) | 8.18 (9.38) | 5.7 (9.39)
  Visit 7 tolerance to 47 celsius heat simulation | 29.28 (25.55) | 32.06 (22.43) | 29.07 (29.28) | 24.85 (26.13)

ADVERSE EVENTS:
Time Frame: The PI will monitor study outcomes. A monthly study staff meeting will be held to review the study progress and discuss any adverse event during study conduction. Adverse event were monitored through study completion, an average of 3 months.
Description: Adverse events will be reported to the PHRC in accordance with the PHRC unanticipated problems including adverse events guidelines. <http://healthcare.partners.org/phsirb/adverse_events.htm>.
Arm/Group | True Acupuncture | Sham Acupuncture | Gabapentin | Sham Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 1/16 | 0/11 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | True Acupuncture (N=15) | Sham Acupuncture (N=16) | Gabapentin (N=11) | Sham Gabapentin (N=14)
Skin Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject participated in a session of sham acupuncture. When the needles, tape, small plastic rings were removed, the acupuncturist noticed redness on the subject's back around the site of the rings. The subject felt no discomfort, itchiness, or pain.

LIMITATIONS AND CAVEATS:
A major limitation is the limited number of study participants in each group. In addition, the use of a sham needle in this pilot study may not have fully differentiated sham versus true electroacupuncture. While the use of diphenhydramine as a placebo control for gabapentin may have mimicked certain side effects of gabapentin, it may have had other confounding effects on the data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT01678586/Prot_SAP_000.pdf